CLINICAL TRIAL: NCT01328730
Title: Post-marketing Study Comparing the Efficacy and Safety of Firebird 2 Versus Cypher Sirolimus-eluting Stents in Treating Patients With Coronary Artery Disease in China
Brief Title: The Real-world Firebird 2 Versus Cypher Sirolimus-eluting Stent in Treating Patients With Coronary Artery Disease
Acronym: REFIRE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: the Cypher SES is now withdrawing in China market
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Cardiovascular Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH20110331
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Stenosis
Keywords: significant stenosis (>70% of lumen stenosis); epicardial coronary arteries.
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Firebird 2 stent group (Experimental): patients who were implated with Firebird 2 SES
  Interventions: Device: Firebird 2 SES
- Cypher Stent Group (Active Comparator): patients who were implanted with Cypher SES
  Interventions: Device: Cypher SES

INTERVENTIONS:
Device: Firebird 2 SES — The FIREBIRD2™ Rapamycin-Eluting CoCr Coronary Stent is the second generation DES of MicroPort, which based on the new cobalt chromium alloy stent platform. It uses polyolefin polymer, which makes the coating property very remarkable.
  Arms: Firebird 2 stent group
Device: Cypher SES — The Cypher SES is based on the 316L platform with Controlled-release, nonresorbable, elastomeric polymer coating.
  Arms: Cypher Stent Group

SUMMARY:
Sirolimus-eluting stent (SES) has been world-widely used in clinical practice in treating patients with coronary artery disease (CAD). The efficacy and safety of Cypher SES (Cordis, MA) has been proved by several randomized clinical trials. Here the investigators design a prospective, multicenter, randomized clinical study in purpose of identifying the non-inferiority in the efficacy and safety in treating CAD patients by Firebird 2 SES (Microport, Shanghai), comparing with Cypher SES.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* male or un-preganant female
* stenosis > 70% in one of major the epicardial coronary arteries
* no contra-indications of stent implantation
* singed the informed consent

Exclusion Criteria:

* acute myocardial infarction within one week
* have contra-indications of stent implantation or can not tolerate dual antiplatelet therapy
* no history of stent implantation within last one-year
* received other brand coronary stent during index procedure
* with no achievement of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
in-stent late lumen loss at 9 months' angiographic follow-up | 9 months
  Late luminal loss was defined as the difference between the minimal luminal diameter immediately after the placement of the stent and the minimal luminal diameter at 9 months

SECONDARY OUTCOMES:
target vessel failure | 1, and 2 years after index procedure
  defined as the occurrence of any of the following within 1 and 2 years after the index procedure: death from cardiac causes, Q-wave or non-Q-wave myocardial infarction, or revascularizationof the target vessel (emergency or elective coronaryartery bypass grafting [CABG] or repeated percutaneous transluminal coronary angioplasty [PTCA]).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China